CLINICAL TRIAL: NCT05852353
Title: Impact, Feasibility, and Acceptability of a Digital Health Intervention for Healthy Children With Pediatric Lower Urinary Tract Symptoms (pLUTS)
Brief Title: Impact, Feasibility, and Acceptability of Bladder Basics
Acronym: Bladder Basics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kathleen Kan, CLINICAL ASSISTANT PROFESSOR, UROLOGY, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 67807; K12DK137162 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-05-10 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Single Group Longitudinal Study looking at pre- and post- results of the same group of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm longitudinal assessment (Experimental): Single arm longitudinal assessment of the feasibility of a digital pediatric bladder health patient education curriculum. The intervention consists of 7 videos that can be viewed over a 4-week time period. Impact on the study objectives will be measured using a longitudinal pre-post intervention study design.
  Interventions: Other: Digital Pediatric Bladder Health Patient Education Curriculum

INTERVENTIONS:
Other: Digital Pediatric Bladder Health Patient Education Curriculum — Bladder Basics is designed to be a digital health intervention to improve knowledge of healthy bladder practices. It is a video-based bladder health curriculum based on 1) principles of Urotherapy 2) stakeholder need for a gold-standard resource 3) behavioral change theory 4) education design standards for inclusion as a comprehensive school health program (CSHP).
  The overall mission of the course is to teach children and their families about pediatric bladder health. The development of the course has followed the NIH's Clear & Simple standards for patient education. The 7 video lesson plan spans 60 minutes total. The course is designed to support families awaiting medical care, which would provide the continued support. In addition, one lesson shares solutions to common home and school-based barriers to behavioral change. The 4 healthy bladder practices that are promoted are- 1) pee every 3 hours 2) drinking water 3) daily poop without straining 4) toilet postures.

SUMMARY:
PLUTS remains a common childhood condition despite effective treatment options. It is important to improve delivery of UT at the clinical level, with future studies that shift pediatric bladder health into a broader community context. This change in contextual setting and scale can impact access to care and disease incidence beyond our current treatment paradigms. Therefore, the overall objective is to measure the early impact and feasibility of a digital health intervention, Bladder Basics. To complete this aim, we will measure clinical and education outcomes pre- and post- intervention and our assessment of acceptability and feasibility will consider framework-based barriers to implementation. Since there is limited existing data with which to build a future intervention, these variables have been carefully considered based on requirements for a future school-based intervention.

DETAILED DESCRIPTION:
The investigators will use a longitudinal pre-post intervention study design to pilot test the acceptability, feasibility, and preliminary educational and clinical outcomes of a novel digital health intervention, Bladder Basics. The primary outcome was the feasibility of recruiting participants to complete BB, which was assessed through metrics on recruitment, engagement, and rates of post-assessment completion. Secondary outcomes included changes in bladder symptoms (both clinical and subjective improvements), bladder health knowledge, and self-efficacy, guided by social cognitive theory. For this pilot study, no control group will be offered. Benefits of this study design include simplicity and ease of administration. As this intervention is virtual, all screening, consent procedures, and study orientation will be conducted using Zoom. Target recruitment numbers will be weighted towards Q2 and Q3 when children are more likely to be in school. The intervention consists of a 7-video curriculum that can be watched on a tablet device, computer, or phone. The videos will be watched in order at the family's convenience within a 4-week period.

Families can pause and restart the course at any time. Their learning progress will be automatically saved and synced across different devices by the online learning platform. The intervention includes 10 activities that include matching, labeling, and revealing hidden information concepts.

Timed surveys with automatic reminders will be administered and stored via a REDCap database. Pre-intervention surveys will be collected prior to obtaining access to the course and will include baseline demographics, knowledge, DVSS, and self-efficacy measures. After watching each lesson, participants will fill out a post-lesson survey to assess their ability to meet the educational objectives which will count as our short-term knowledge measure. After watching the entire course, participants will have up to 4 weeks from the start of the course to complete the first post-intervention survey. This will include a repeat measure of DVSS and self-efficacy, as well as a new assessment of acceptability, education design, and open-ended feedback questions on perceived structural barriers to adopting bladder health practices and areas for program improvement. A second post-intervention survey will be distributed at 3-months from the start of the course (long-term), and will include a repeat measure of DVSS and knowledge of bladder health practices. The time difference in measuring educational and clinical outcomes reflect the theory that the investigators would expect some degree of time to transpire between knowledge acquisition and repeated practices leading to subjective improvement. Screening, consent, study orientation procedures, and RedCap database management will be managed by a research assistant consistent with prior studies. The investigator will conduct the descriptive and quantitative data analysis portion of the study. Quantitative analysis will be performed using SPSS. The primary investigator will lead overall study completion and address any study-related obstacles or concerns. Alternative approaches include qualitative analysis of open-ended feedback questions using an iterative team-based approach to thematic analysis with myself, 1 research assistant, and 1 medical student who have both been previously trained in this method.

Expected outcomes: The investigators hypothesize that this study will demonstrate that Bladder Basics is a feasible and acceptable program for families facing pLUTS. The investigators expect robust study recruitment based on prior community interest and studies. Information obtained for this study will be used to 1) improve our existing intervention to help families awaiting pLUTS care and 2) design a school-based intervention. Data from this proposal will be submitted for presentation at academic conferences and to relevant journals for manuscript publication.

ELIGIBILITY:
Inclusion Criteria:

* Parents or guardians >= 18 years of age
* involved in the care of a child 5-10 years old with bladder problems
* English speaking

Exclusion Criteria:

* Individuals <18 years old.
* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Liu C, Chu J, Hughes T, Follis C, Kan KM. Empowering Bladder Health Education for Children: Integrating Situated Learning Theory and the ARCS Model in Online Program Design. J Pediatr Health Care. 2026 Jan-Feb;40(1):112-127. doi: 10.1016/j.pedhc.2025.09.005. Epub 2025 Oct 9. PMID 41065601
- [Result] Liu C, Chu J, Kan KM. Effectiveness of an Online Health Education Program for Pediatric Lower Urinary Tract Symptoms. Urology. 2025 Oct;204:171-178. doi: 10.1016/j.urology.2025.05.058. Epub 2025 May 31. PMID 40456454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents of children aged 5-10 years with presence of lower urinary tract symptoms (LUTS), defined as dysfunctional voiding scoring system (DVSS) score > 6 for girls, >9 for boys, were recruited from our pediatric urology clinic, local pediatric practices and the community. Community recruitment involved flyers posted in public libraries, community and childcare centers and community-based organizations.
Pre-assignment Details: 268 families met eligibility criteria. 15 families submitted surveys the were found to be fraudulent. 102 families signed informed consent and were assigned to the study arm.
Groups:
- Single Arm Longitudinal Assessment: Each family (parent-child dyad) receives the intervention (digital pediatric bladder health patient education curriculum). The intervention consists of 7 videos that can be viewed over a time period of up to 4 weeks.
Period: Overall Study
Arm/Group | Single Arm Longitudinal Assessment
Started (Includes 102 parents and 102 children.) | 102
Signed informed consent (child with LUTS) (Includes 72 parents and 72 children.) | 72
Signed informed consent (child did not have LUTS) (Includes 30 parents and 30 children.) | 30
Completed intervention (child with LUTS) (Includes 52 parents and 52 children.) | 52
Completed intervention (child did not have LUTS) (Includes 23 parents and 23 children.) | 23
Completed 4-week survey (child with LUTS) (Includes 51 parents and 51 children.) | 51
Completed 4-week survey (child did not have LUTS) (Includes 23 parents and 23 children.) | 23
Completed 12-week survey (child with LUTS) (Includes 47 parents and 47 children.) | 47
Completed 12-week survey (child did not have LUTS) (Includes 21 parents and 21 children.) | 21
Completed (Includes 68 parents and 68 children.) | 68
Not Completed | 34
Not completed — Family (dyad with LUTS) who consented but withdrew | 2
Not completed — Family (dyad did not have LUTS) who consented but withdrew | 1
Not completed — Family (dyad) who consented but did not complete intervention | 24
Not completed — Family (dyad) who completed intervention but was lost to follow-up | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed the intervention, and in which the child in the dyad had presence of lower urinary tract symptoms at baseline (DVSS score > 6 in girls, > 9 in boys)
Groups:
- Parent-Child Dyad - Parent Participants; Parent-Child Dyad - Child Participants: Each parent-child dyad receives the intervention (digital pediatric bladder health patient education curriculum). The intervention consists of 7 videos that can be viewed over a time period of up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Parent-Child Dyad - Parent Participants | Parent-Child Dyad - Child Participants | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 70 | 70
  Between 18 and 65 years | 70 | 0 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 47 | 111
  Male | 6 | 23 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or European, not Hispanic or Latino | 33 | 37 | 70
  Asian or Asian American, not Hispanic or Latino | 27 | 21 | 48
  Hispanic or Latino/a | 8 | 7 | 15
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American, not Hispanic or Latino | 1 | 1 | 2
  Middle Eastern or North African | 1 | 1 | 2
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Recruited
Description: Recruitment was measured as the number and percentage of individuals who expressed interest, were screened, and provided consent.
Time Frame: 3 months
Population: Parent-child dyads who completed the screening survey.
Measure: Count of Participants; unit: Participants
Groups:
- Parent-Child Dyad: Each family (parent-child dyad) receives the intervention (digital pediatric bladder health patient education curriculum). The intervention consists of 7 videos that can be viewed over a time period of up to 4 weeks.
Arm/Group | Parent-Child Dyad
Number analyzed (Participants) | 429
Participants
  Expressed Interest (submitted survey) - all dyads | 429
  Eligible for Participation - dyads with LUTS at baseline | 183
  Consented - dyads with LUTS at baseline, excludes withdrawn dyads | 70

2. Primary Outcome: Engagement: Video Completion Rate
Description: Engagement was measured by assessing the video completion rate (videos watched/total videos) as calculated by the video platform.
Time Frame: 3 months
Population: Parent-child dyads who signed informed consent, did not withdraw, and in which the child in the dyad had presence of lower urinary tract symptoms at baseline (DVSS score > 6 in girls, > 9 in boys)
Measure: Count of Participants; unit: Participants
Arm/Group | Parent-Child Dyad
Number analyzed (Participants) | 70
Participants
  Completed 80% - 100% of the curriculum | 50
  Completed 20% - 80% of the curriculum | 2
  Completed 0% - 20% of the curriculum | 18

3. Primary Outcome: Post-assessment Completion Rates
Description: Post-assessment completion was measured as the percentage of participants who completed surveys following the Bladder Basics videos. After completing the videos, participants completed surveys to test knowledge, and collect data regarding user feedback and symptom improvement. The 2 post-intervention surveys were sent at 4-weeks and 12-weeks post-baseline.
Time Frame: 4-weeks and 12-weeks
Population: Parent-child dyads who completed the Bladder Basics video (based on parent's self-report) and completed initial post-lesson survey, and in which the child in the dyad had presence of lower urinary tract symptoms at baseline (DVSS score > 6 in girls, > 9 in boys)
Measure: Count of Participants; unit: Participants
Arm/Group | Parent-Child Dyad
Number analyzed (Participants) | 52
Participants
  Completed 4-week survey | 51
  Completed 12-week survey | 47

4. Secondary Outcome: Change in Dysfunctional Voiding Symptom Score (DVSS) to Evaluate Bladder Health Clinical Outcomes
Description: To evaluate the impact of Bladder Basics on short- and long-term bladder health clinical outcomes by comparing baseline and post-intervention Dysfunctional Voiding Symptom Score (DVSS) questionnaire results in healthy children ages 5-10 years old with pediatric lower urinary tract symptoms. The survey consists of 10 questions, each scored from 0 to 3 (0 = Almost Never; 1 = Less Than Half the Time; 2 = About Half the Time; 3 = Almost Every Time). Scores were summed to create the overall score (0 to 30). Children with a higher DVSS score have more frequent symptoms and/or behavioral problems
Time Frame: baseline, 4-weeks; 12-weeks
Population: Children with LUTS at baseline and who completed the 4-week and 12-week surveys, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Child Group: Children aged 5-10 years with LUTS.
Arm/Group | Child Group
Number analyzed (Participants) | 51
score on a scale
  baseline score - 4-week survey completers (both genders) | 11.51 (3.12)
  4-weeks score - 4-week survey completers (both genders) | 8.47 (4.61)
  baseline score - 4-week survey completers (girls): number analyzed (Participants) | 37
  baseline score - 4-week survey completers (girls) | 11.38 (3.41)
  4-weeks score - 4-week survey completers (girls): number analyzed (Participants) | 37
  4-weeks score - 4-week survey completers (girls) | 8.30 (4.37)
  baseline score - 4-week survey completers (boys): number analyzed (Participants) | 14
  baseline score - 4-week survey completers (boys) | 11.86 (2.25)
  4-weeks score - 4-week survey completers (boys): number analyzed (Participants) | 14
  4-weeks score - 4-week survey completers (boys) | 8.93 (5.34)
  baseline score - 12-week survey completers (both genders): number analyzed (Participants) | 47
  baseline score - 12-week survey completers (both genders) | 11.53 (3.17)
  12-weeks score - 12-week survey completers (both genders): number analyzed (Participants) | 47
  12-weeks score - 12-week survey completers (both genders) | 6.62 (3.87)
  baseline score - 12-week survey completers (girls): number analyzed (Participants) | 35
  baseline score - 12-week survey completers (girls) | 11.40 (3.43)
  12-weeks score - 12-week survey completers (girls): number analyzed (Participants) | 35
  12-weeks score - 12-week survey completers (girls) | 6.80 (3.95)
  baseline score - 12-week survey completers (boys): number analyzed (Participants) | 12
  baseline score - 12-week survey completers (boys) | 11.92 (2.35)
  12-weeks score - 12-week survey completers (boys): number analyzed (Participants) | 12
  12-weeks score - 12-week survey completers (boys) | 6.08 (3.73)

5. Secondary Outcome: Pre-intervention to Post-intervention Knowledge Survey Created by ResearchTeam
Description: To evaluate the impact of Bladder Basics on improving knowledge of pediatric bladder health practices by comparing baseline pre-intervention to post-intervention survey results in parents of healthy children ages 5-10 years old with pediatric lower urinary tract symptoms. Knowledge surveys will be created by study team. The survey consists of 11 questions. Correct answers are scored as 1, incorrect answers are scored as 0. Question scores were summed to create an overall score of 0 to 11, with higher scores corresponding to better knowledge about bladder health.
Time Frame: Baseline, Post-lesson (approximately 4 weeks) and 12 weeks post-intervention
Population: Parents of children with LUTS at baseline and who completed immediate post-video survey and 12-week survey, respectively.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Parent Group: Parent/legal guardians of children aged 5-10 years with LUTS.
Arm/Group | Parent Group
Number analyzed (Participants) | 52
score on a scale
  Baseline - post-lesson survey completers | 10 [9 to 11]
  Post-lesson score - post-lesson survey completers | 11 [10.25 to 11]
  Baseline - 12-week survey completers: number analyzed (Participants) | 47
  Baseline - 12-week survey completers | 10 [9 to 11]
  12-week score - 12-week survey completers: number analyzed (Participants) | 47
  12-week score - 12-week survey completers | 11 [11 to 11]

6. Secondary Outcome: Validated Self-efficacy Survey
Description: To measure the acceptability and feasibility of the Bladder Basics education program.
  The self-efficacy survey is adapted from Parents Patient Activation Measure-13 (PPAM-13). Participants answered questions as strongly disagree, disagree, agree, strongly agree, and NA. Raw scores were transformed to an overall scale of 0 to 100. Higher scores indicate higher levels of self-efficacy.
Time Frame: Baseline and 4 weeks
Population: Parents of children with LUTS at baseline and who completed the baseline and 4-week surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Group
Number analyzed (Participants) | 51
score on a scale
  Baseline | 63.12 (16.82)
  4-weeks | 70.84 (17.16)

7. Secondary Outcome: Validated Acceptability Survey
Description: To measure the acceptability and feasibility of the Bladder Basics education program.
  The acceptability survey is developed based on the Technology Acceptance Theory. The survey contains 13 questions assessing perceived usefulness, perceived ease of use, attitude towards intervention, and behavioral intention for future use. Each question is assessed on a 5-point Likert scale, each with a range from 1 (strongly disagree) to 5 (strongly agree). Scores are summed and averaged to create the overall score, with a range of 1 to 5 (higher scores indicate better acceptability).
Time Frame: Immediately after completing the videos (up to 4 weeks following baseline)
Population: Parents of children with LUTS at baseline who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Group
Number analyzed (Participants) | 52
score on a scale | 4.306 (0.490)

8. Secondary Outcome: Validated Education Design Survey -- Parents
Description: To measure the acceptability and feasibility of the Bladder Basics education program.
  This survey is adapted from the Attention, Relevance, Confidence, and Satisfaction (ARCS) questionnaire. Each question is scored on a 5-point Likert scale ranging from 1 (not true) to 5 (very true). Scores are summed and averaged to create overall score (range: 1 to 5). Higher scores indicate better education design.
Time Frame: Immediately after completing the videos (up to 4 weeks following baseline)
Population: Parents of children with LUTS at baseline who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Group
Number analyzed (Participants) | 52
score on a scale | 4.31 (0.49)

9. Secondary Outcome: Validated Education Design Survey - Children
Description: To measure the acceptability and feasibility of the Bladder Basics education program.
  This survey is adapted from the Attention, Relevance, Confidence, and Satisfaction (ARCS) questionnaire. Each question is scored on a 5-point Likert scale ranging from 1 (not true) to 5 (very true).
Time Frame: Immediately after completing the videos (up to 4 weeks following baseline)
Population: Children with LUTS at baseline who completed the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Child Group
Number analyzed (Participants) | 52
Participants
  Fun: Strongly disagree | 1
  Fun: Disagree | 1
  Fun: Neither agree or disagree | 4
  Fun: Agree | 15
  Fun: Strongly agree | 31
  Important: Strongly disagree | 1
  Important: Disagree | 1
  Important: Neither agree or disagree | 2
  Important: Agree | 12
  Important: Strongly agree | 36
  Easy: Strongly disagree | 0
  Easy: Disagree | 1
  Easy: Neither agree or disagree | 7
  Easy: Agree | 20
  Easy: Strongly agree | 24
  Enjoyable: Strongly disagree | 3
  Enjoyable: Disagree | 1
  Enjoyable: Neither agree or disagree | 2
  Enjoyable: Agree | 16
  Enjoyable: Strongly agree | 30

10. Secondary Outcome: Open-ended Feedback Questions to Measure Acceptability and Feasibility of Education Program
Description: Number of excerpted items obtained from participant feedback according to topic area.
  To measure acceptability and feasibility of Bladder Basics with consideration of stakeholder, educational design, and behavioral change theory barriers.
  Open-ended feedback questions were used to characterize the intervention's ability to be used as a population-level intervention. Feedback was coded according to topic area.
Time Frame: Immediately after completing the videos (up to 4 weeks following baseline)
Population: The Overall Number of Participants Analyzed represents the number of parent-child dyads who completed the Bladder Basics video (based on parent's self-report) and who completed initial post-intervention survey, and in which the child in the dyad had presence of lower urinary tract symptoms at baseline (DVSS score > 6 in girls, > 9 in boys).
Measure: Count of Units; unit: Excerpts
Units Other Than Participants: Excerpts
Arm/Group | Parent-Child Dyad
Number analyzed (Participants) | 52
Number analyzed (Excerpts) | 312
Excerpts
  Affective attitude | 48
  Age appropriateness | 10
  Burden | 90
  Course content: Educational topics | 15
  Course content: Presentation format | 43
  Future content: Epidemiology of pediatric bladder health | 3
  Future content: Bathroom use best practices | 8
  Future content: Bathroom pathology content | 28
  Future content: Dietary Information and Bowel habits | 9
  Future content: Format suggestions | 10
  Future content: No changes needed | 24
  General acceptability | 6
  Intervention coherence | 6
  Perceived effectiveness | 12

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Parent-Child Dyad - Parent Participants | Parent-Child Dyad - Child Participants
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05852353/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT05852353/SAP_002.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05852353/ICF_000.pdf